CLINICAL TRIAL: NCT01069796
Title: A Multi Phase II Clinical Trials Evaluating the Association of Bevacizumab With Weekly Paclitaxel and Capecitabine in First Line Treatment for Patients With Triple Negative Metastatic or Locally Advanced Cancer
Brief Title: Bevacizumab + Paclitaxel + Capecitabine in Triple Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The number of inclusion was reached normally
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-Taxel (GINECO BR108)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Triple Negative Metastatic Breast Cancer
Keywords: triple negative; metastatic; breast cancer; First line chemotherapy
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms | interventions — Paclitaxel; Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Association bevacizumab paclitaxel capecitabine breast cancer (Experimental): * bevacizumab 10 mg/kg in IV, D1 and D15
  * paclitaxel 80mg/m2 in IV, D1 to D8 and D15
  * capecitabine 1600mg/m2/D, per os, D1 to D5, Weeks 1,2 and 3
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m² weekly
Drug: Bevacizumab — 10 mg/kg d1 d15
Drug: Capecitabine — 800 mg/m² p.o. twice a day, D1 to D5 week 1, 2 & 3

SUMMARY:
Patients with triple negative metastatic breast cancer (HER2-, PR-, ER-) will receive bevacizumab, paclitaxel and capecitabine as a first line of treatment (possibility to have received adjuvant chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Female histologically confirmed adenocarcinoma of the breast ER-, PR-, HER2- disease
* Measurable disease
* Patients may received prior radiotherapy as adjuvant treatment or/and metastatic disease provided that they have progressive disease at study entry

Exclusion Criteria:

* Prior chemotherapy for metastatic disease
* HER2 positive and/or hormonal receptor positive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
objective response rate | 36 months for recrutment and 30 months for follow up

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Centre Paul Papin, Angers
  - Clinique Tivoli, Bordeaux
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre Hospitalier Intercommunal, Fréjus
  - Clinique des 4 Pavillons, Lormont
  - Hôpital Privé Clairval, Marseille
  - Centre Azuréen de Cancérologie, Mougins
  - Centre Alexis Vautrin, Nancy
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Régional, Orléans
  - Institut Jean Godinot, Reims
  - Hôpitaux Drôme Nord - Site de Romans-sur-Isère, Romans-sur-Isère
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Clinique de l'Union, St.-Jean
  - Centre Paul Strauss, Strasbourg
  - Centre Hospitalier Bretagne Atlantique, Vannes